CLINICAL TRIAL: NCT01177150
Title: A First-in-Human Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Escalating Oral Doses of JNJ 28431754 in Healthy Male Subjects
Brief Title: A First-in-Human Study of JNJ-28431754 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Study Physician, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR012454; 28431754NAP1001
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Sodium-Glucose Transporter 2; Canagliflozin; Pharmacodynamic; Pharmacokinetic; Safety; Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 001 (Experimental): JNJ-28431754/ Placebo Part 1: One oral dose of JNJ 28431754 (10 mg to 600 mg) or matching placebo will be administered after an overnight fast of at least 10 hours .For patients who receive a previously tested dose as 2 equally divided doses the evening dose will be administered at 10 hours after the morning dose.
  Interventions: Drug: JNJ-28431754/ Placebo
- 002 (Experimental): JNJ-28431754 Part 2: A single dose of JNJ-28431754 will be orally administered on 2 occasions (14 days apart) after an overnight fast of at least 10 hours with and without a standard meal.
  Interventions: Drug: JNJ-28431754

INTERVENTIONS:
Drug: JNJ-28431754/ Placebo — Part 1: One oral dose of JNJ 28431754 (10 mg to 600 mg) or matching placebo will be administered after an overnight fast of at least 10 hours .For patients who receive a previously tested dose as 2 equally divided doses, the evening dose will be administered at 10 hours after the morning dose.
  Arms: 001
Drug: JNJ-28431754 — Part 2: A single dose of JNJ-28431754 will be orally administered on 2 occasions (14 days apart) after an overnight fast of at least 10 hours with and without a standard meal.
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and or the pharmacodynamics (PD) of single oral doses of JNJ-28431754 in healthy male volunteers. The study will evaluate the PK and PD effects of study drug in volunteers who fasted compared to those who did not fast before study drug administration.

DETAILED DESCRIPTION:
This is a single-center study that will be conducted in two Parts (Part 1 and Part 2). Volunteers may participate in Part 1 or Part 2 of the study but not in both Part 1 and Part 2. Part 1 of the study will evaluate the safety and tolerability of single, oral (by mouth) escalating (increasing) doses of JNJ 28431754 (ranging from 10 mg to 600 mg) or placebo in healthy male volunteers. The pharmacokinetics (PK), how JNJ 28431754 is absorbed, distributed, and removed from the body over time and pharmacodynamics (PD), the effects JNJ-28431754 has on the body, will also be evaluated. Part 2 of the study is a randomized, 2 period crossover study where 8 eligible male volunteers will receive a single oral dose of JNJ 28431754 on 2 occasions (14 days apart) with and without food (ie, a standard meal) to assess the effect of co-administration with food on the PK and PD of JNJ-28431754. In Part 1, at least 48 healthy male volunteers who meet entry criteria will be randomized (assigned by chance) into 6 cohorts (dose groups) and receive a single oral dose of study drug (JNJ-28431754 or placebo); study drug will be assigned to volunteers double-blinded (neither the investigator or the volunteer will know the identity of the assigned treatment). One or more additional cohorts may be added to the study; the additional cohort may test a previously tested dose of JNJ 28431754 as 2 equally divided doses, to be administered 10 hours apart. Each volunteer will participate in one dose group only. Each dose group will evaluate a different dose strength of JNJ-28431754 (10 mg to 600 mg) starting at the lowest dose. Volunteers in each dose group will be required to stay overnight in the clinical research unit (CRU) for 6 nights to receive study drug and to have safety, tolerability, PK, and PD assessments performed. Patients will return to the CRU for a final safety follow-up visit 10 to 14 days after study drug administration. For each volunteer, the total duration of Part 1 of the study will be at least 5 weeks (includes a 3-week screening period). In Part 2 of the study, 8 eligible male volunteers will receive a single oral dose of JNJ 28431754 on 2 occasions (14 days apart) with and without food (ie, a standard meal); JNJ-28431754 will be administered to volunteers as "open-label" treatment (ie, volunteers will know that they are receiving active drug) . Part 2 will begin after sufficient data has been collected from Part 1 to select the dose of JNJ-28431754 for Part 2 of the study (the dose selected will be within the dose range evaluated in Part 1 of the study). Volunteers will be required to stay overnight in the CRU for 5 nights on 2 occasions to receive study drug and to have post dose safety, tolerability, PK, and PD assessments performed. Patients will return to the CRU for a final safety follow-up visit 10 to 14 days after the 2nd single-dose administration of JNJ-38431754. For each volunteer, the total duration of Part 2 of the study will be approximately 7 weeks (includes a 3-week screening period and about a 2-week interval between the 2 single-dose administrations of JNJ 38431754). Volunteers in Part 1 and Part 2 of the study will be monitored for safety during the study by evaluating adverse events reported and results from vital signs measurements, electrocardiograms, physical examinations performed and laboratory tests. Part 1: One dose of JNJ-28431754 (10mg to 600mg) or placebo will be administered after an overnight fast of at least 10 hours (for additional cohorts, previously tested doses will be administered as 2 equally divided doses taken 10 hours apart). Part 2: One dose of JNJ-28431754 will be administered on 2 occasions (14 days apart) after an overnight fast of at least 10 hours with and without a standard meal. All doses of study drug will be administered to patients orally using an oral dispenser.

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index (BMI) between 20.0 and 29.9 kg/m2 inclusive
* Be a non-smoker or non-tobacco user (not smoked cigarettes or used tobacco-containing products for at least 6 months prior to screening)
* Have competency in speaking and comprehending the language where the study will be conducted

Exclusion Criteria:

* Have history, or family history of bleeding or coagulation disorders or history of disorders that are potential causes of occult (test positive for fecal blood test without visible blood in feces) gastrointestinal bleeding
* Have currently active skin disorders
* Have history of renal or urinary tract diseases
* Have history of having chronically taken (daily administration for more than 7 days) oral steroids, topical iodine, aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), anticoagulants or other drugs known to interfere with blood clotting within 3 months of study start, or anticipates a need to take any of these during the course of the study
* Have history of recent major surgery (within 6 months of study start)
* Have history of recent travel (within 6 months) to locations that may predispose to the acquisition of communicable illnesses (e.g., parasitic or water-borne illnesses in developing tropical regions)
* Have recent history of alcohol or drug abuse within 6 months prior to screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by evaluating adverse events reported and results from vital signs measurements, electrocardiograms, physical examinations performed and laboratory tests. | From Screening (within 21 days prior to Day 1) up to Day 14 or at the time of early withdrawal

SECONDARY OUTCOMES:
Urine Glucose Excretion (the amount of glucose excreted in the urine per 24 hours and the amount of glucose excreted in each urine collection fraction) | At protocol-specified timepoints before and after study drug administration on Day 1
The renal threshold for Urinary Glucose Excretion | At protocol-specified timepoints before and after study drug administration on Day 1
Plasma glucose, serum insulin and serum C peptide concentrations measured from blood samples collected | At protocol-specified timepoints before and after study drug administration on Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.